CLINICAL TRIAL: NCT01736982
Title: Contingency Management for Smoking Cessation in the Homeless
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-186-2; R21DA031897 (NIH)
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Cigarette Smoking
Keywords: Cigarette Smoking; Homeless; Contingency Management; Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): transdermal nicotine replacement [21 mg patches (4 wks), 14 mg (2 wks), 7 mg (2 wks)], breath sample monitoring, standard smoking cessation counseling
  Interventions: Other: Standard of Care
- Standard of Care plus Contingency Management (Experimental): Standard smoking cessation intervention plus contingency management
  Interventions: Behavioral: Contingency Management; Other: Standard of Care

INTERVENTIONS:
Behavioral: Contingency Management — Participants earn reinforcement in the form of prizes for breath samples that test negative for cigarette smoking.
  Arms: Standard of Care plus Contingency Management
Other: Standard of Care — Standard smoking cessation counseling
Other: Standard of Care — transdermal nicotine replacement [21 mg patches (4 wks), 14 mg (2 wks), 7 mg (2 wks)]
Other: Standard of Care — Breath sample monitoring

SUMMARY:
Smoking cessation services are an unmet need among the homeless, who smoke at rates more than 3 times the national estimate; successful interventions in this underserved population have the potential for improving individual and public health. Contingency management (CM) is a behavioral intervention with efficacy in a number of substance use disorder populations, including smokers. However, no known studies have evaluated the effect of CM in homeless smokers. The investigators plan to examine smoking-related outcomes in homeless treatment-seeking smokers (N = 70) randomized to standard care smoking cessation (transdermal nicotine replacement therapy [NRT] + standard counseling + carbon monoxide [CO] monitoring) or standard care plus CM (NRT + standard counseling + CO monitoring + CM) conditions. Standard counseling and CO monitoring will occur for the first 4 weeks, with NRT use continuing through week 8. Participants in both conditions will meet with study staff up to twice daily on weekdays for biochemical verification of smoking status. Participants in the CM condition will have the opportunity to earn prizes for negative breath samples (CO ≤ 4 ppm) up to twice daily on weekdays. CO breath samples will be collected at all visits. The investigators expect that participants randomized to CM will have better outcomes compared to those in standard care.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* homeless
* regular smoker

Exclusion Criteria:

* non-English speaking
* contra-indications for transdermal nicotine
* in recovery for pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Longest Duration of Abstinence | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Carla J Rash, PhD, Principal Investigator — UConn Health
Locations (1):
- The Friendship Center, New Britain, Connecticut, United States